CLINICAL TRIAL: NCT06493578
Title: A Randomized, Double-Blind, Vehicle-Controlled Phase 2b Trial Evaluating the Efficacy, Safety & Pharmacokinetics of VYN201 Gel in the Treatment of Non Segmental Vitiligo
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of VYN201 Gel in Subjects With Non-segmental Vitiligo.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VY2024-02
Record Dates: First submitted 2024-03-18; First posted 2024-07-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Non-segmental Vitiligo
Keywords: NSV; VYN201 Gel; vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, double-blind, vehicle-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose VYN201 (1.0%) (Active Comparator): Subjects will apply VYN201 1.0% once daily on affected vitiligo areas. The first part of the study will be a 24-week, double-blind, vehicle controlled treatment period. Following, the second part will be a 28-week, double-blind treatment extension period, with a 4-week safety follow-up period after the last investigational medicinal product (IMP) dose. After completion of the Week 24 assessments, subjects randomized to 1.0% will remain and continue on the same dose until Week 52.
  Interventions: Drug: VYN201 Gel
- Mid dose VYN201 (2.0%) (Active Comparator): Subjects will apply VYN201 2.0% once daily on affected vitiligo areas. The first part of the study will be a 24-week, double-blind, vehicle controlled treatment period. Following, the second part will be a 28-week, double-blind treatment extension period, with a 4-week safety follow-up period after the last investigational medicinal product (IMP) dose. After completion of the Week 24 assessments, subjects randomized to 2.0% will remain and continue on the same dose until Week 52.
  Interventions: Drug: VYN201 Gel
- High dose VYN201 (3.0%) (Active Comparator): Subjects will apply VYN201 3.0% once daily on affected vitiligo areas. The first part of the study will be a 24-week, double-blind, vehicle controlled treatment period. Following, the second part will be a 28-week, double-blind treatment extension period, with a 4-week safety follow-up period after the last investigational medicinal product (IMP) dose. After completion of the Week 24 assessments, subjects randomized to 3.0% will remain and continue on the same dose until Week 52.
  Interventions: Drug: VYN201 Gel
- Vehicle (Placebo Comparator): Subjects will apply VYN201 vehicle (placebo) once daily on affected vitiligo areas. The first part of the study will be a 24-week, double-blind, vehicle controlled treatment period. Following, the second part will be a 28-week, double-blind treatment extension period, with a 4-week safety follow-up period after the last investigational medicinal product (IMP) dose. After completion of the Week 24 assessments, subjects randomized to vehicle (placebo) will be re-randomized to 1 of the 3 higher VYN201 (active) dose groups (1.0%, 2.0% or 3.0% once daily) in a 1:1:1 ratio while maintaining the blind until Week 52.
  Interventions: Drug: VYN201 Gel; Drug: Vehicle Gel

INTERVENTIONS:
Drug: VYN201 Gel — VYN201 Gel is a topical formulation applied as a thin layer to affected areas.
Drug: Vehicle Gel — Vehicle gel (placebo) is matching in appearance to VYN201 gel and is to be applied in the same manner as VYN201 gel.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of VYN201 Gel in subjects with non-segmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed and signed an Informed Consent Form (ICF) prior to any study-related procedures.
2. Able to understand and comply with study requirements.
3. Male or female aged 18 to 75 years, inclusive.
4. Clinical diagnosis of non-segmental vitiligo where the total affected BSA does not exceed 10%.
5. F-VASI score of ≥0.5 and ≤3.0.
6. T-VASI score of ≥3.0 and ≤10.0.
7. Agree to discontinue all agents used to treat vitiligo from Screening through the study completion. Over-the-counter preparations deemed acceptable by the investigator are permitted.
8. If receiving concomitant medication for any reason other than vitiligo, must be on a stable regimen at Screening, and anticipating staying on a stable regimen through the study completion.
9. Female participants must:

   * Be of non-childbearing potential (i.e., surgically sterilized [hysterectomy, bilateral salpingectomy, bilateral oophorectomy, tubal ligation/occlusion at least 6 weeks before the Screening]) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause) OR
   * If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception from signing the ICF until at least 1 month after the last dose of IMP. An acceptable method of contraception includes one of the following:

     1. Hormonal contraception (for at least 3 months prior to Screening) in combination with a barrier method.
     2. Intrauterine device (placement at least 3 months prior to Screening).
     3. Diaphragm with spermicide.
     4. Cervical cap with spermicide.
     5. Condoms with spermicide.
     6. Vasectomized partner (6 months minimum since vasectomy).
10. Male participants, if not biologically or surgically sterilized, must agree not to donate sperm and, if engaging in sexual intercourse, must agree to use a condom from signing the ICF until at least 1 month after the last dose of study drug. If engaging with a female partner who could become pregnant, the female partner must additionally use an acceptable method of contraception for this same period.

Exclusion Criteria:

1. Clinical diagnosis of other forms of vitiligo (e.g., segmental) or other hypo- or de-pigmentation skin diseases (e.g., piebaldism, leukoderma, Vogt-Koyanagi-Harada disease, malignancy induced hypopigmentation, etc.).
2. Concomitant dermatologic conditions or other medical condition(s) which may, in the opinion of the investigator, interfere with IMP application or study assessments.
3. History of melanocyte transplantation procedure or depigmentation treatment [e.g. Monobenzyl ether of hydroquinone (Monobenzone)].
4. Visible test site skin injury, damage, or observations in or around the application site which, in the opinion of the investigator, will interfere with study assessments or increase participation risk.
5. Dyed hair in the treatment area that could interfere with any clinical assessments.
6. Significant facial hair or are unable to maintain very short cropped facial hair (<5mm) during course of the study.
7. Leukotrichia in >33% of vitiligo lesional surface of the face or the body.
8. History or presence of any clinically significant condition(s) which, in the opinion of the investigator, could interfere with the course of the study or expose the participant to undue risk by participating in this study, including, but not limited to: metabolic, allergic, cardiovascular, pulmonary, hepatic, renal, hematologic (including bleeding disorders), gastrointestinal (including peptic ulcer disease, gastritis or bleeding diathesis, excluding appendectomy or hernia repair), endocrine, immunologic, dermatologic, muscular, neurological, psychiatric, neoplastic, or other disease(s).
9. Major surgery within 3 months of randomization or with planned major surgery during trial.
10. Current or recent history (<30 days before Screening and/or <45 days before randomization) of a clinically meaningful bacterial, fungal, parasitic, or mycobacterial infection.
11. Any known or suspected premalignant or malignant disease within 5 years prior to Screening (excluding successfully treated basal or squamous cell carcinomas, actinic keratoses, melanoma in situ, cervical dysplasias, cervical cancer).
12. Systemic biologic or immune-modulating treatment within 12 weeks prior to Screening and through study completion or topical treatment in the vitiligo areas within 2 weeks prior to Screening and through study completion.
13. Received any investigational therapy, device or procedure within 30 days or 5 half-lives (whichever is longer) prior to Screening. Investigational biologics should be discussed with the sponsor to determine if a longer period of discontinuation is required.
14. Relevant (in the investigator opinion) ultraviolet light exposure including phototherapy within 8 weeks prior to Screening.
15. Use of any other prior and concomitant therapy not listed above that, in the opinion of the investigator, may interfere with the evaluation of study outcomes, including drugs that cause photosensitivity or skin pigmentation (e.g. antibiotics such as tetracyclines, antifungals). These medications should be discontinued within 4 weeks of randomization.
16. Known or suspected history of alcohol or drug abuse within 12 months of Screening or in the opinion of the investigator, will interfere with the subject's ability to comply with the administration schedule and study assessments (alcohol abuse is defined as regular consumption of >10 standard units of alcohol per week).
17. Subjects who are pregnant or breastfeeding.
18. Clinically significant abnormal laboratory values at Screening:

    1. Neutrophils < lower limit of normal.
    2. Hemoglobin < 10 g/dL.
    3. Platelets < 100 × 109/L.
    4. Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 2.0 × upper limit of normal.
    5. Estimated creatinine clearance < 30 mL/min or renal disease requiring dialysis as determined by Cockcroft-Gault.
    6. Positive serology tests for Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), or human immunodeficiency virus (HIV)-1 and HIV-2 antibody.
19. Subjects who received a live vaccine within 4 weeks prior to Screening.
20. Subjects with known allergy or reaction to any component of the study formulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of VYN201 compared to vehicle at Week 24 in subjects with NSV. | Week 24
  Proportion of subjects who achieve a ≥50% improvement from Baseline in F-VASI score at Week 24.

SECONDARY OUTCOMES:
To evaluate the efficacy of VYN201 as measured by F-VASI over time in subjects with NSV. | Week 24 and Week 52
  Mean and percent changes from Baseline in F-VASI at Week 24 and Week 52.
To evaluate the efficacy of VYN201 as measured by T-VASI assessment over time in subjects with NSV. | Week 52
  Proportion of subjects who achieve a ≥50% improvement from baseline in T-VASI at Week 52

OTHER OUTCOMES:
To evaluate the efficacy of VYN201 as measured by T-VASI assessment over time in subjects with NSV. | Week 24 and Week 52
  Mean and percent changes from Baseline in T-VASI at Week 24 and Week 52.
To evaluate the efficacy of VYN201 as measured by Vitiligo Noticeability Scale over time in subjects with NSV. | Week 52
  Vitiligo Noticeability Scale (VNS) is the subjects' perception of their vitiligo. A rating of 'More noticeable' would indicate the subject perceived the treatment as ineffective and a rating of 'No longer noticeable' would indicate the subjects' perceived the treatment to be highly effective.
  The assessment is rated by the following measures:
  1. More noticeable
  2. As noticeable
  3. Slightly less noticeable
  4. A lot less noticeable
  5. No longer noticeable
To evaluate the efficacy of VYN201 as measured by T-VASI assessment over time in subjects with NSV. | Week 24
  Proportion of subjects who achieve a ≥50% improvement from baseline in T-VASI at Week 24.
To evaluate the safety and tolerability of VYN201 as measured by Treatment-Emergent Adverse Events (TEAEs) over time in subjects with NSV. | Baseline through Week 56
  Frequency and severity of TEAEs. TEAEs will be defined as events that emerge after the first application of IMP having been absent pre-treatment, or worsens relative to the pre-treatment state.
To evaluate the safety and tolerability of VYN201 as measured by Physical Examinations over time in subjects with NSV. | Baseline through Week 56
  Changes from baseline in physical examination findings.
  General physical examinations will include: height (cm) and weight (kg), head and neck, eyes, ears, nose and throat, lymph nodes, and the cardiovascular, respiratory systems, abdominal, urologic, and musculoskeletal systems.
  Targeted physical examinations will be a symptom-directed evaluation and will include body weight and assessment(s) of the body systems or organs, as indicated by subject's symptoms, AEs, or other findings.
To evaluate the safety and tolerability of VYN201 as measured by ECGs over time in subjects with NSV. | Baseline through Week 56
  Changes from baseline in ECG assessments. A standard 12-lead ECG will be used to obtain RR interval (ms), PR interval (ms), QRS interval (ms), QT interval (ms), QTcF (ms), and QTcB (ms).
To evaluate the efficacy of VYN201 as measured by vital signs over time in subjects with NSV. | Baseline through Week 56
  Changes from baseline of vital signs. The following will be monitored as safety variables:
  * Systolic and diastolic blood pressure (mmHg)
  * Pulse rate (beats per minute)
  * Respiration rate (breaths per minute)
  * Arterial oxygen saturation (SpO2)
  * Body temperature (°C)
To evaluate the efficacy of VYN201 as measured by Laboratory Tests over time in subjects with NSV. | Baseline through Week 56
  Changes from baseline in Laboratory Safety assessments. Assessed laboratory values include the following: clinical chemistry/biochemistry, hematology, coagulation parameters, urinalysis, urine drug screen, and viral serology.
To evaluate the safety and tolerability of VYN201 as measured by Local Skin Tolerability assessment over time in subjects with NSV. | Baseline through Week 56
  Changes from baseline in Local Skin Tolerability. Assessment of the dryness, scaling, erythema, hyperpigmentation, burning/stinging and pruritus of the affected area. Incidence of severity grades in skin tolerability are assessed with the following severity scoring:
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe
To determine the PK of VYN201 in subjects with NSV (Dose Proportionality) | Week 24 and Week 52
  Dose response relationship with VYN201
To determine the PK of VYN201 in subjects with NSV (Time to Steady State Ratio) | Week 24 and Week 52
  Time to Steady State Ratio
To determine the PK of VYN201 in subjects with NSV (Cmax) | Baseline through Week 52
  Maximum observed plasma concentration of VYN201
To determine the PK of VYN201 in subjects with NSV (Accumulation Ratio) | Week 24 and Week 52
  Ratio of VYN201 accumulation under steady state conditions
To determine the PK of VYN201 in subjects with NSV (Tmax) | Baseline through Week 52
  Time to reach Maximum observed plasma concentration of VYN201

CONTACTS AND LOCATIONS:
Locations (49):
- United States (42):
  - Cahaba Dermatology & Skin Health Center, Birmingham, Alabama
  - Saguaro Dermatology, Phoenix, Arizona
  - Center for Dermatology and Plastic Surgery/CCT Research, Scottsdale, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Clinical Trial Institute of Northwest Arkansas, LLC, Fayetteville, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology Research, Inc, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - Marvel Clinical Research, Huntington Beach, California
  - Northridge Clinical Trials, Northridge, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Integrative Skin Science and Research, Sacramento, California
  - Clarity Dermatology, Castle Rock, Colorado
  - Colorado Medical Research Center, Denver, Colorado
  - Skin Care Research, Boca Raton, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Skin Care Research, Hollywood, Florida
  - International Clinical Research - FL LLC, Sanford, Florida
  - Metabolic Research Institute, Inc, West Palm Beach, Florida
  - MetroMed Clinical Trials, Chicago, Illinois
  - DS Research of Southern Indiana, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research of Kentucky, Louisville, Kentucky
  - DelRicht Research at Audubon Dermatology, New Orleans, Louisiana
  - Lawrence J. Green, MD LLC, Rockville, Maryland
  - JDR Dermatology Research, Las Vegas, Nevada
  - The Skin Center Dermatology Group, New City, New York
  - Bobby Buka MD, PC, New York, New York
  - Hickory Dermatology Research Center, Hickory, North Carolina
  - The Skin Surgery Center for Clinical Research, Winston-Salem, North Carolina
  - Clarity Dermatology, Canal Winchester, Ohio
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Cumberland Skin Center for Clinical Research, Hermitage, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Newco 3A Research, El Paso, Texas
  - Center for Clinical Studies, LTD.LLP, Houston, Texas
  - Austin Insitute for Clinical Research, Pflugerville, Texas
  - DelRicht Research at Lockhart Matter Dermatology, Prosper, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
- Canada (7):
  - Dermatology Research Institute, Calgary, Alberta
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - JRB Research Inc, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Research Toronto, Toronto, Ontario
  - Siena Medical Research, Montreal, Quebec